CLINICAL TRIAL: NCT00028535
Title: Phase I Trial of Interleukin-12 in Combination With Paclitaxel Plus Herceptin in Patients With Her2-positive Malignancies
Brief Title: Interleukin-12, Paclitaxel, and Trastuzumab in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01407; 1999C0326; OSU-0167; NCI-84; OSU-99H0326; CDR0000069102; U01CA076576 (NIH)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Recurrent Endometrial Carcinoma; Recurrent Gastric Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma | interventions — Trastuzumab; Paclitaxel; Taxes; Interleukin-12 Subunit p35; Interleukin-12

ARMS (1):
- Arm I (Experimental): Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15 and paclitaxel IV over 3 hours on day 1 of course 1. Beginning with course 2, patients receive trastuzumab and paclitaxel as in course 1 and interleukin-12 subcutaneously on days 2, 5, 9, 12, 16, and 19. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: paclitaxel; Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: recombinant interleukin-12 — Given SC
  Other Names: cytotoxic lymphocyte maturation factor; IL-12; interleukin-12; natural killer cell stimulatory factor; Ro 24-7472

SUMMARY:
Phase I trial to study the effectiveness of interleukin-12, paclitaxel, and trastuzumab in treating patients who have solid tumors. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining interleukin-12, chemotherapy, and monoclonal antibody therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of interleukin-12 when given in combination with paclitaxel and trastuzumab (Herceptin®) in patients with HER2/neu-overexpressing malignancies.

II. Determine the response rate and time to progression in patients treated with this regimen.

III. Determine the anti-tumor effect of this regimen in these patients.

OUTLINE: This is a dose-escalation study of interleukin-12.

Patients receive trastuzumab (Herceptin®) IV over 30-90 minutes on days 1, 8, and 15 and paclitaxel IV over 3 hours on day 1 of course 1. Beginning with course 2, patients receive trastuzumab and paclitaxel as in course 1 and interleukin-12 subcutaneously on days 2, 5, 9, 12, 16, and 19. Courses repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of interleukin-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2/neu-overexpressing (2+ or 3+) malignancy by any standardized assay (fluorescence in-situ hybridization allowed)
* Measurable or evaluable disease
* Failed standard curative therapy
* No brain or CNS metastasis
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - Karnofsky 70-100%
* At least 6 months
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 8 g/dL (transfusion or epoetin alfa allowed)
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3.0 times ULN
* Hepatitis B surface antigen negative
* Creatinine no greater than 1.5 times ULN
* Calcium no greater than 11 mg/dL (calcium-lowering agents allowed)
* No active or unstable cardiovascular disease
* No cardiac disease requiring drug or device intervention
* No coronary artery disease
* No congestive heart failure
* Cardiac ejection fraction normal by echocardiogram or MUGA scan
* No significant peripheral neuropathy
* No significant CNS disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No serious concurrent infection requiring IV antibiotic therapy
* No clinically significant autoimmune disease (e.g., rheumatoid arthritis)
* No clinically significant gastrointestinal bleeding
* No uncontrolled peptic ulcer disease
* No inflammatory bowel disease
* No other major illness that would preclude study participation
* No other concurrent malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix
* No prior interleukin-12
* No prior trastuzumab (Herceptin®)
* At least 3 weeks since prior chemotherapy
* At least 3 weeks since prior hormonal therapy
* No concurrent systemic corticosteroids
* At least 3 weeks since prior radiotherapy
* At least 3 weeks since prior surgery
* At least 3 weeks since prior investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-11; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
MTD of IL-12, defined as the dose level one level beneath that dose at which 2 or more of 6 patients showed DLT, based on the NCI CTC version 2.0 | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States